CLINICAL TRIAL: NCT05048498
Title: An Open Pilot Study to Assess the Pharmacokinetics, Tolerability, and Safety of NEX-18a Given as a Subcutaneous Injection for the Treatment of Intermediate 2 or Higher-risk MDS, CMML or AML
Brief Title: Pharmacokinetics, Tolerability and Safety of NEX-18a
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanexa AB (Industry)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NEX-18-01
Record Dates: First submitted 2021-05-11; First posted 2021-09-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Myelodysplastic Syndromes (MDS); Chronic Myelomonocytic Leukemia (CMML); Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azacitidine (Active Comparator): Treatment phase 1: the patients will receive regular treatment with azacitidine for 4 days.
  Treatment phase 2: the patients will receive regular treatment with azacitidine for 3 days.
  Interventions: Drug: Azacitidine Injection
- NEX-18a (Experimental): Treatment phase 1: the azacitidine dose for day 5 will be replaced by a single dose NEX-18a
  Treatment phase 2: the azacitidine dose for day 4 and 5 will be replaced by a single dose NEX-18a
  Interventions: Drug: NEX-18a injection

INTERVENTIONS:
Drug: NEX-18a injection — In Treatment phase 1, NEX-18a will be given as a single subcutaneous injection.
  In Treatment phase 2, NEX-18a will be given as a single subcutaneous injection.
  Other Names: PharmaShell; Azacitidine; 5-azacitidine
  Arms: NEX-18a
Drug: Azacitidine Injection — In Treatment phase 1, azacitidine will be administered once daily for four days. In Treatment phase 2, azacitidine will be administered once daily for three days.
  Other Names: Azacitidine; 5-azacitidine; Vidaza
  Arms: Azacitidine

SUMMARY:
The study will evaluate the safety, tolerability and pharmacokinetics of NEX-18a, a long-acting injectable azacitidine, in patients diagnosed with intermediate 2 or higher-risk MDS, CMML, or AML and already on treatment with azacitidine.

DETAILED DESCRIPTION:
Since 2010, subcutaneous treatment with azacitidine has been the first-line treatment for patients with high-risk MDS. Azacitidine has been established as a standard of care and is described in the National Comprehensive Cancer Network (NCCN) guidelines as a core component of optimal treatment of MDS. However, mainly due to its short half-life (41 minutes) when administered subcutaneously azacitidine should, according to the approved label, be administered for seven consecutive days at a dose of 75 mg/m2 body surface area (BSA) each 28-day cycle. In the Nordic Guidelines, two alternative dosing schedules may also be considered: 100 mg/m2 BSA sc day 1-5 or 75 mg/m2 BSA sc day 1-5 + 8-9 (to avoid injection during weekends).

Nanexa AB has developed NEX-18a, a subcutaneous injection of azacitidine with extended-release based on the drug delivery system, PharmaShell®. Drug particles are enclosed in a coating with controlled solubility, and as the coating dissolves over time the drug is released in a predefined manner. This technique provides a way to create drugs with a prolonged release for parenteral administration. The technology used by Nanexa to manufacture the coating is via Atomic Layer Deposition (ALD). In ALD, reactive gases are used which build up a surface coating with high precision, atomic layer by atomic layer.

NEX-18a will offer a benefit to current azacitidine treatment with a reduction of subcutaneous administrations, decreased need for pre-medication, and will reduce the time each patient has to spend in the hospital in order to receive the treatment in each cycle. In addition, the patients will spend less time traveling to and from the hospital and from a health care perspective, one injection instead of seven per cycle will reduce the time and the resources the health care provider dedicates to treating the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to any study specific procedures.
2. Female and male patients ≥ 18 years of age.
3. Body Mass Index (BMI) > 19 and < 30 kg/m2 BSA at screening.
4. Treatment with azacitidine corresponding to 100 mg/m2 BSA x 5 per treatment cycle for at least six cycles for:

   1. intermediate-2 and high-risk myelodysplastic syndromes (MDS) according to the International Prognostic Scoring System (IPSS)
   2. chronic myelomonocytic leukemia (CMML) with 10-29 % marrow blasts
   3. acute myeloid leukemia (AML) according to World Health Organization (WHO) classification
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
6. Recovery of Hematology and Clin. Chemistry assessment according to clinical praxis at the start of the last azacitidine treatment cycle before the screening visit.
7. Female subject must be of non-childbearing potential (defined as pre-menopausal females with a documented tubal ligation or hysterectomy or bilateral oophorectomy; or as post-menopausal females defined as 12 months' amenorrhoea [in questionable cases a blood sample with simultaneous follicle stimulation hormone 25-140 IE/L and estradiol < 200 pmol/L is confirmatory])
8. Male patients must agree to use an adequate method of contraception. Male patients who are sexually active must use, with their partner, a condom AND one of the following methods of highly effective contraception from the time of IMP administration until 90 days after the last dose of IMP.

   1. oral (except low-dose gestagen (lynestrenol and norestisteron)), injectable or implanted hormonal contraceptives
   2. intrauterine device
   3. intrauterine system (for example progestin-releasing coil)
   4. vasectomized male (with appropriate post vasectomy documentation of the absence of sperm in the ejaculate)
   5. bilateral tubal occlusion or hysterectomy
9. Willingness and ability to comply with study procedures, visit schedules, study restrictions, and requirements.

Exclusion Criteria:

1. The patient has participated in any other investigational/interventional trial including an investigational drug within 30 days (or five half-lives of the study drug prior to screening, whichever is longer) prior to screening.
2. Diagnosis of malignant disease within the previous 5 years (excluding basal cell carcinoma of the skin without complications, "in-situ" carcinoma of the cervix or breast, or other local malignancy excised or irradiated with a high probability of cure).
3. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from participating in the study.
4. The patient has a history of alcohol abuse or drug abuse within the past 12 months.
5. Any condition including the presence of laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study.
6. Lack of suitability for participation in the study, for any reason, judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Hematology and Clinical Chemistry analyses | 0-30 days
  Change from baseline to 30 days follow-up. Descriptive individual data.
Adverse events | 0-30 days
  Change from baseline to 30 days follow-up. Descriptive individual data.
Vital signs | 0-30 days
  Change from baseline to 30 days follow-up. Descriptive individual data.
Physical examination | 0-30 days
  Change from baseline to 30 days follow-up. Descriptive individual data.
Local tolerance (injection site) | 0-30 days
  Change from baseline to 30 days follow-up. Descriptive individual data.
Concomitant medications/therapy | 0-30 days
  Change from baseline to 30 days follow-up. Descriptive individual data.

SECONDARY OUTCOMES:
AUC-time curve | 0-24 h
  From time 0 to 24 hours
AUC from time 0-last | 0-336 h
  From time 0 to last
AUC from time 0 to infinity | 0-336 h
  From time 0 to infinity
Plasma Concentration | 0-336 h
  Maximum Plasma Concentration
Plasma Concentration over time | 0-336 h
  Plasma Concentration at 336h
Half-life measurement | 0-336 h
  Terminal elimination half-life
Measurement of distribution | 0-336 h
  Volume of distribution
Elimination | 0-336 h
  Clearance
Local tolerance of NEX-18a | 0-30 days
  Change from baseline to 30 days follow-up. Descriptive individual data. The local tolerance will be measured by inspection of injection sites. Pain, tenderness erythema/redness, and induration/swelling will be assessed by a four-grade scale where 1 is mild and 4 is potentially life threatening.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Olsson Strömberg, MD, Principal Investigator — Uppsala University, Uppsala, Sweden
Locations (2):
- Sweden (2):
  - Karolinska University Hospital Huddinge, Huddinge
  - Kliniska Forsknings och Utvecklings Enheten KFUE, Uppsala

IPD SHARING:
Plan to Share IPD: No